CLINICAL TRIAL: NCT00657124
Title: Preoperative Oral Supplementation of Carbohydrate and Branched-Chain Amino Acids-Enriched Nutrient Improves Insulin Resistance in Patients With Hepatectomy; Prospective Randomized Clinical Trial by Using Artificial Pancreas
Brief Title: Effect of Preoperative Supplementation in Insulin Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kochi University (Other)
Responsible Party: Kochi Medical School, Kochi University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PEA-AP-01; Kochi University
Record Dates: First submitted 2008-04-07; First posted 2008-04-14 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Liver Disease
Keywords: AEN
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): receive a preoperative supplementation with carbohydrate and branched-chain amino acids-enriched nutrient
  Interventions: Dietary Supplement: Aminolevan EN
- 2 (Placebo Comparator): receive a preoperative supplementation without carbohydrate and branched-chain amino acids-enriched nutrient
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aminolevan EN — The present study used carbohydrate and BCAA-enriched soft-powder nutrient-mixture for preoperative supplementation. Supplementation with Aminolevan EN (100 g per day) started at two weeks prior to the surgery under the careful monitoring of compliance.
  Arms: 1
Dietary Supplement: Placebo — placebo
  Other Names: No receive, normal diet
  Arms: 2

SUMMARY:
To elucidate the effect of preoperative supplementation of carbohydrate and branched-chain amino acids on postoperative insulin resistance in patients undergoing hepatic resection, we set a randomized trial.

DETAILED DESCRIPTION:
Twenty-six patients with hepatectomy due to a live tumor were prospectively randomized to receive a preoperative supplementation with carbohydrate and branched-chain amino acids-enriched nutrient or not.

ELIGIBILITY:
Inclusion Criteria:

* The present study employed 26 patients, who underwent elective liver resection for hepatocellular carcinoma or adenocarcinoma.

Exclusion Criteria:

* body weight loss greater than 10 per cent during 6 months prior to the surgery
* distant metastasis
* or seriously impaired function of vital organs due to respiratory, renal or heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
to evaluate the total amount of insulin required for glycemic control after hepatic resection | total amount of insulin required

SECONDARY OUTCOMES:
to investigate the trends of postoperative blood glucose levels and the incidence of severe hypoglycemia (< 40 mg/dL) by using artificial pancreas during intensive care unit stay | hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Takehiro Okabayashi, MD, Study Director — Kochi Medical School, Kochi University
Locations (1):
- Kochi Medical School, Nankoku, Kohasu-Okocho, Japan